CLINICAL TRIAL: NCT02220543
Title: The Effectiveness of a Biopsychosocial Rehabilitation Program in Primary Care (Back on Track) Versus Primary Care as Usual in Patients With Chronic Low Back Pain in Which Psychosocial Factors Minimally Influence Daily Life Functioning: a Randomized Controlled Trial
Brief Title: Chronic Low Back Pain Rehabilitation in Primary Care: an RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Adelante, Centre of Expertise in Rehabilitation and Audiology (Other); The Province of Limburg (Unknown); CZ Fonds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-3-019
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain; Chronic Pain; Musculoskeletal Pain
Keywords: Cognitive behavioral therapy; Primary health care; Physical Therapy
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Musculoskeletal Pain | interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Back on Track intervention (Experimental): Back on Track intervention is a biopsychosocial primary care intervention
  Interventions: Other: Back on Track intervention; Other: Primary care as usual
- Primary care as usual (Active Comparator): Primary care as usual comprises maximally 12 individual regular physical therapy sessions for a maximum of 8 weeks.
  Interventions: Other: Back on Track intervention; Other: Primary care as usual

INTERVENTIONS:
Other: Back on Track intervention — Biopsychosocial primary care intervention based on multidisciplinary pain rehabiliation programs. The Back on Track intervention comprises 4 individual sessions and 8 group sessions.
Other: Primary care as usual — Regular physical therapy in primary care. Physical therapists are recommended by their profession (the Royal Dutch Society for Physical Therapy) to work according to a profession-specific guideline for the treatment of patients with low back pain in primary care settings. Maximally 12 individual sessions (30 minutes each) for a maximum of 8 weeks.

SUMMARY:
The aim of this study is to evaluate the effectiveness and cost-effectiveness of a new primary care intervention "Back on Track" as compared to usual primary care in patients with non-specific chronic low back pain in which disability levels are moderate and the role of psychosocial factors to this disability is at maximum low (classified as WPN2).

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain; defined as pain between scapulae and gluteal region, whether or not with radiation towards one or both legs, present for at least three months.
* Presence of contributing social and psychological factors, however not complex (WPN2 classification)
* Age between 18 and 65 year
* Sufficient knowledge of the Dutch language
* Acceptance towards the biopsychosocial approach instead of biomedical approach

Exclusion Criteria:

* Chronic low back pain attributable to e.g. infection, tumour, osteoporosis, fracture, structural deformation, inflammatory process, radicular syndrome or cauda equina syndrome
* Pregnancy
* Any suspicion of an (underlying) psychiatric disease, for which psychiatric treatment is better suited, according to the expert opinion of the consultant in rehabilitation medicine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Quebec Back Pain Disability Scale (QBPDS) | Change in functional disability between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
  The QBPDS is a 20-itemed questionnaire designed to determine the individuals' functional disability level (ranging from 0-100). A higher score reflects higher disability.

SECONDARY OUTCOMES:
Credibility and Expectancy Questionnaire (CEQ) | Directly after the first treatment (in the first week of the intervention)
EuroQol-5D (EQ-5D) | Change in quality of life between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Hospital Anxiety and Depression Scale (HADS) | Change in anxiety and depression between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Pain Catastrophizing Scale (PCS) | Change in catastrophizing between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Numeric Rating Scale (NRS) | Change in pain intensity between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Tampa Scale of Kinesiophobia | Change in kinesiophobia between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Pain Self-Efficacy Questionnaire (PSEQ) | Change in self-efficacy between pre-treatment (baseline) and post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Global Perceived Effect (GPE) | Global perceived effect at post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up
Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TiC-P) | Medical consumption at pre-treatment (baseline), post-treatment (with an expected average of 8 weeks), 3 months follow-up and 12 months follow-up after the end of the treatment
Social demographic questionnaire | pre-treatment
Treatment questionnaire | Post-treatment (with an expected average of 8 weeks)
  This questionnaire contains only one question and asks patients directly after the treatment program has finished (post-treatment) to indicate whether they think they have received the new intervention or care as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan PJ Huijnen, Dr., Principal Investigator — Maastricht University
Locations (8):
- Netherlands (8):
  - Fysiotherapie Giessen-Ploemen, Bunde, Limburg
  - Fysiohof, Maastricht, Limburg
  - Fysio Zuyd Caberg, Maastricht, Limburg
  - Fysiotherapiepraktijk Yvonne Janss, Maastricht, Limburg
  - ICM Fysio, Maastricht, Limburg
  - Fysiotherapie Breuers, Margraten, Limburg
  - Fysiotherapie Abbink, Ulestraten, Limburg
  - Fysio Valkenburg, Valkenburg, Limburg

REFERENCES:
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Lindstrom I, Ohlund C, Eek C, Wallin L, Peterson LE, Fordyce WE, Nachemson AL. The effect of graded activity on patients with subacute low back pain: a randomized prospective clinical study with an operant-conditioning behavioral approach. Phys Ther. 1992 Apr;72(4):279-90; discussion 291-3. doi: 10.1093/ptj/72.4.279. PMID 1533941
- [Background] Leeuw M, Goossens MEJB, van Breukelen GJP, de Jong JR, Heuts PHTG, Smeets RJEM, Koke AJA, Vlaeyen JWS. Exposure in vivo versus operant graded activity in chronic low back pain patients: results of a randomized controlled trial. Pain. 2008 Aug 15;138(1):192-207. doi: 10.1016/j.pain.2007.12.009. Epub 2008 Feb 1. PMID 18242858
- [Background] Lamb SE, Hansen Z, Lall R, Castelnuovo E, Withers EJ, Nichols V, Potter R, Underwood MR; Back Skills Training Trial investigators. Group cognitive behavioural treatment for low-back pain in primary care: a randomised controlled trial and cost-effectiveness analysis. Lancet. 2010 Mar 13;375(9718):916-23. doi: 10.1016/S0140-6736(09)62164-4. Epub 2010 Feb 25. PMID 20189241
- [Background] Macedo LG, Smeets RJ, Maher CG, Latimer J, McAuley JH. Graded activity and graded exposure for persistent nonspecific low back pain: a systematic review. Phys Ther. 2010 Jun;90(6):860-79. doi: 10.2522/ptj.20090303. Epub 2010 Apr 15. PMID 20395306
- [Background] Brunner E, De Herdt A, Minguet P, Baldew SS, Probst M. Can cognitive behavioural therapy based strategies be integrated into physiotherapy for the prevention of chronic low back pain? A systematic review. Disabil Rehabil. 2013 Jan;35(1):1-10. doi: 10.3109/09638288.2012.683848. Epub 2012 May 21. PMID 22607157
- [Derived] van Erp RMA, Huijnen IPJ, Koke AJA, Abbink FE, den Hollander M, Smeets RJEM. Development and content of the biopsychosocial primary care intervention 'Back on Track' for a subgroup of people with chronic low back pain. Physiotherapy. 2017 Jun;103(2):160-166. doi: 10.1016/j.physio.2016.04.004. Epub 2016 May 11. PMID 27641497
- [Derived] van Erp RM, Huijnen IP, Verbunt JA, Smeets RJ. A biopsychosocial primary care intervention (Back on Track) versus primary care as usual in a subgroup of people with chronic low back pain: protocol for a randomised, controlled trial. J Physiother. 2015 Jul;61(3):155. doi: 10.1016/j.jphys.2015.03.003. Epub 2015 Apr 23. PMID 25922158